CLINICAL TRIAL: NCT03587987
Title: Manikin Study of the Comparison of Two Different Resuscitation Devices (Neopuff and rPAP) During Simulated Resuscitation in the Neonatal Unit
Brief Title: Comparison of Two Different Resuscitation Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Dr. Gene Dempsey, Principal Investigator, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ECM 4 (x) 05/06/18
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Manual Ventilation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neopuff (Active Comparator): neopuff
  Interventions: Device: Neopff
- r PAP (Experimental): rPap device
  Interventions: Device: rPap

INTERVENTIONS:
Device: Neopff — manual ventilation
  Arms: Neopuff
Device: rPap — Manual ventilation
  Arms: r PAP

SUMMARY:
There is a complex physiological process involved in establishing regular breaths at birth. After initiation of the first breath, fluid is removed from the alveoli and enough pressure must be generated to inflate the lungs . Most newborns will establish spontaneous regular breathing sufficient to maintain the heart rate above 100 beats/min and to improve perfusion within 3 minutes of birth. According to the neonatal resuscitation programme (NRP), if heart rate is below 100 or there is persistence of apnoea or gasping after the initial steps of drying/stimulation and oropharyngeal suction, intervention is required .

The main focus of neonatal resuscitation is effective ventilation to improve gas exchange and prevent respiratory failure. After birth, approximately 4% to 10% of term and late preterm newborns will receive help breathing with positive-pressure ventilation (PPV). Adequate mask ventilation is essential when providing breaths during neonatal resuscitation. However, this can be difficult, especially for less experienced staff and may be affected by inadequate seal of the mask, gas leaks and airway obstruction. In addition, trauma may be caused by the volumes being given during pressure controlled ventilation.

DETAILED DESCRIPTION:
Comparison of two different neonatal resuscitation devices (Neopuff and rPAP) in the Neonatal Unit in Cork University Maternity Hospital. Participants will use the devices on a mannequin. Performance of the two devices is judged by comparing the tidal volumes produced.

Participants will be recruited from the medical staff (Non-consultant Hospital Doctors and Consultants) of the neonatal unit.

ELIGIBILITY:
Inclusion Criteria:

1. Neonatology consultants and NCHD's from CUMH
2. Participants must have completed Neonatal Resuscitation Programme (NRP)
3. Participants must be working as doctors in the area of neonatology

Exclusion Criteria:

1. Any history of cardiac or respiratory disorder
2. Physicians who are post-call

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Percentage difference in expired tidal volumes produced by rPAP versus Neopuff resuscitation devices during simulated resuscitation using neonatal mannequins | 1 minutre

CONTACTS AND LOCATIONS:
Locations (1):
- UCC, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No